CLINICAL TRIAL: NCT02739880
Title: Evaluation of the Effect of Multi-point Intra-mucosal Injections of Cross-linked Hyaluronic Acid (DESIRIAL®) in the Vaginal Vestibule: A Prospective, Bicentric, Pilot Study
Brief Title: Multi-point Intra-mucosal Injections of Cross-linked Hyaluronic Acid (DESIRIAL®) in the Vaginal Vestibule
Acronym: INREG 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Laboratoires Vivacy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2016/PM-001; 2016-A00124-47 (Other: ANSM)
Record Dates: First submitted 2016-04-06; First posted 2016-04-15 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2019-03

CONDITIONS: Menopause; Dyspareunia
Keywords: Vaginal discomfort; Vaginal dryness
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The study population (Experimental): The study population consists of postmenopausal patients (more than 2 years and less than 10 years) with a body mass index <35 with sexual disorders (dyspareunia) or vaginal discomfort associated with vaginal dryness.
  Intervention: Intra-mucosal Injections of Cross-linked Hyaluronic Acid
  Interventions: Device: DESIRIAL® (Intra-mucosal Injections of Cross-linked Hyaluronic Acid)

INTERVENTIONS:
Device: DESIRIAL® (Intra-mucosal Injections of Cross-linked Hyaluronic Acid) — Multi-point Intra-mucosal Injections of Cross-linked Hyaluronic Acid (DESIRIAL®) in the Vaginal Vestibule
  The intervention is Intended for intra-mucosal injection in women for biostimulation / rehydration of the surface layers of the lining of the genital areas, vaginal hypotrophies and / or treatment of female sexual dysfunction related to subsidence G "spot or area of Gräfenberg ".
  Following disinfection and topical anesthesia (lidocaine gel), the vesitbule is injected using a multi-point technique. The optimal volume of DESIRIAL® to be used for injection into the vestibule is approximately 0.3 ml in total.
  Other Names: Cross-linked Hyaluronic Acid; DESIRIAL®

SUMMARY:
The main objective of this study is to measure changes in the thickness of the vaginal lining (epithelium + underlying stroma) between 0 and 8 weeks after injection.

DETAILED DESCRIPTION:
The secondary objectives of this study are to measure changes in the following between 0 and 8 weeks after injection:

A. vaginal flora and Nugent score.

B. vaginal pH.

C. functional evolution via the VHI index by Gloria Bachman (state of the vaginal mucosa), pain / dyspareunia (visual analog scale) and the satisfaction concerning care viay the PGI-I questionnaire (Patient Global Impression and Improvement).

D. Procollagen I and III gene expression (by PCR) and mitotic activity of the mucosa (Ki67 proliferation marker) based on biopsies.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 8 weeks of follow-up
* The patient is menopausal (amenorrhea) for over 2 years and less than 10 years
* The patient has a body mass index <35
* The patient has sexual disorders (dyspareunia) or vaginal discomfort associated with vaginal dryness.

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant or breastfeeding
* The patient is not menopausal (both clinically and biologically)
* The patient has a body mass index > 35
* The patient has a genital prolapse higher than stage 2 with a surgical indication
* The patient has stress incontinence with a surgical indication
* The patient suffers from vaginismus
* Presence of an untreated viral, fungal or bacterial vulvovaginal or urinary infection
* Hemorrhagic or neoplastic genital pathologies
* Existence of a hormone-dependent tumor, genital bleeding of unknown origin
* Current treatments based on antihypertensives, steroid anti-inflammatory drugs, anticoagulants, major antidepressants, aspirin
* Known hypersensitivity to hyaluronic acid or mannitol
* Known hypersensitivity to Betadine
* Known hypersensitivity to Lidocaine
* Hypersensitivity to EMLA®
* Previous urogynaecological vulvovaginal surgery

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
The thickness of the vaginal mucosa on a histological section | Day 0
The thickness of the vaginal mucosa on a histological section | Week 8

SECONDARY OUTCOMES:
Vaginal pH | Day 0
Vaginal pH | Week 8
Vaginal flora (on Pap smear) | Day 0
Vaginal flora (on Pap smear) | Week 8
Nugent score (on Pap smear) | Day 0
Nugent score (on Pap smear) | Week 8
PGI-I (Patient Global Impression and Improvement) Questionnaire | Week 8
The Vaginal Health Index by Gloria Bachman | Day 0
The Vaginal Health Index by Gloria Bachman | Week 8
Pain (dyspareunia) by visual analog scale | Day 0
Pain (dyspareunia) by visual analog scale | Week 8
Measurement of collagen expression (procollagen I and III) | Day 0
Measurement of collagen expression (procollagen I and III) | Week 8
Level of Ki67 proliferation marker | Day 0
Level of Ki67 proliferation marker | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Berreni, MD, Study Director — Centre Médical Karis
Locations (2):
- France (2):
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - Centre Médical KARIS, Perpignan

REFERENCES:
- [Result] Berreni N, Salerno J, Chevalier T, Alonso S, Mares P. Evaluation of the effect of multipoint intra-mucosal vaginal injection of a specific cross-linked hyaluronic acid for vulvovaginal atrophy: a prospective bi-centric pilot study. BMC Womens Health. 2021 Aug 28;21(1):322. doi: 10.1186/s12905-021-01435-w. PMID 34454465